CLINICAL TRIAL: NCT00178724
Title: Spinal Cord Injury Registry - North American Clinical Trials Network for Spinal Cord Injury
Brief Title: Spinal Cord Injury Registry - North American Clinical Trials Network
Acronym: NACTN
Status: Recruiting | Type: Observational
Sponsor: Robert G. Grossman, MD (Other)
Collaborators: Christopher Reeve Paralysis Foundation (Other); The Methodist Hospital Research Institute (Other); The University of Texas Health Science Center, Houston (Other); University of Virginia (Other); University of Louisville (Other); University of Toronto (Other); University of Maryland, Baltimore (Other); Walter Reed National Military Medical Center (U.S. Federal Agency); Thomas Jefferson University (Other); University of Miami (Other); Brooke Army Medical Center (U.S. Federal Agency); Louisiana State University Health Sciences Center in New Orleans (Other); Vanderbilt University Medical Center (Other); Medical College of Wisconsin (Other); Duke University (Other)
Responsible Party: Sponsor-Investigator, Robert G. Grossman, MD, Professor, Department of Neurosurgery, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Other Study IDs: Pro00002187; W81XWH-16-C-0031 (Other Grant/Funding Number: Department of Defense); CTN16-2020(RG) (Other: NACTN)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; SCI; traumatic spinal cord injury; acute spinal cord injury; paralysis
MeSH Terms: conditions — Spinal Cord Injuries; Paralysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Treatment Given: Any male or female 18 years or older admitted to a NACTN hospital, at the time of injury, with an initial (first time) spinal cord injury caused by trauma and has paralysis (muscle weakness) or loss of sensation (touch). The patient has not received medical or surgical care for this injury prior to admission to a NACTN hospital. Patient or family member must give consent to participate.
  Interventions: Other: No Treatment Given

INTERVENTIONS:
Other: No Treatment Given — Intervention is not given.

SUMMARY:
The NACTN Spinal Cord Injury Registry is a network of clinical centers collecting de-identified data from patients admitted through the Emergency Department of a NACTN center at the time of injury with an initial (first time) spinal cord injury (SCI). Information will be collected on the natural history of SCI and course of treatment through the first 12 months from the date of injury or long as medically indicated. Data collected includes imaging information from CT or MRI scans, neurological and general medical outcome and rehabilitation evaluation. No intervention is given other than standard of care for spinal cord injury, intensive monitoring and frequent follow up care.

DETAILED DESCRIPTION:
The participating centers include:

University of Texas Health Science Center, Houston; University of Toronto, Toronto; University of Virginia, Charlottesville; University of Louisville, Louisville; University of Maryland, Baltimore; Walter Reed National Military Medical Center, Bethesda; Thomas Jefferson University, Philadelphia; University of Miami, Miami; Brooke Army Medical Center, Fort Sam Houston; Louisiana State University Health Sciences Center, New Orleans; Vanderbilt University Medical Center, Nashville; Medical College Wisconsin, Milwaukee; Duke University, Durham

The NACTN Clinical Coordinating Center is located at:

Houston Methodist Hospital, Houston

The Center for Biostatistics is located at:

Houston Methodist Hospital, Houston

The Data Management Center is located at:

University of Louisville, Louisville

Preliminary work has been completed on the selection of data elements, data collection protocols, case record form design, and the design of a computer system for clinical data management and data quality control.

In the first phase of the network, data will be collected on the natural history of SCI. Although there is considerable data in the literature about the natural history of SCI, current changes in treatment appear to be modifying the natural history. In particular very early surgery, including decompression of the spinal cord and vertebral stabilization with instrumentation appears, in some cases of SCI, to be improving outcomes.

No treatment is given other than standard of care for SCI. Data is collected in hopes to help SCI patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Any patient male or female > or equal to 18 years of age with first time spinal cord injury caused by trauma and has neurological deficit with paralysis (weakness) or loss of sensation (touch).
* Has not received prior medical of surgical care for this injury at an intermediate hospital.
* Must give informed consent

Exclusion Criteria:

* Any patient or family refusing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted to a NACTN hospital through the Emergency Department at the time of injury.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2005-07; Primary Completion 2025-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
International Standards For Neurological Classification of Spinal Injury (ISNCSCI) | Pre-operative, Post-operative, 2 weeks, Discharge, 3 months, 6 months, 12 months, 36 months and 48 months
  A neurological assessment and classification of a spinal cord injury

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Grossman, MD, Study Chair — Houston Methodist Hospital, Houston; Karl M Schmitt, MD, Principal Investigator — The University of Texas, Houston; Michael G Fehlings, MD, PhD, Principal Investigator — University of Toronto/Toronto Western Hospital, Toronto; Emily Sieg, MD, Principal Investigator — University of Louisville, Louisville; Bizhan Aarabi, MD, Principal Investigator — University of Maryland Medical Center, Baltimore Shock Trauma Center; Chun-Po Yen, MD, Principal Investigator — University of Virginia Health System, Charlottesville; Christopher J Neal, MD, Principal Investigator — Walter Reed National Military Medical Center, Bethesda; James S Harrop, MD, Principal Investigator — Thomas Jefferson University, Philadelphia; James D Guest, MD, PhD, Principal Investigator — University of Miami, Miami; Ryan P Morton, MD, Principal Investigator — Brooke Army Medical Center, Fort Sam Houston; Jason D Wilson, MD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans; Hamid Shah, MD, Principal Investigator — Vanderbilt University Medical Center, Nashville; Shekar N Kurpad, MD, PhD, Principal Investigator — Medical College of Wisconsin, Milwaukee; Christopher I Shaffrey, MD, Principal Investigator — Duke University, Durham
Locations (14):
- United States (13):
  - University of Miami, Miami, Florida
  - University of Louisville Health Sciences Center, Louisville, Kentucky
  - Louisiana State University Medical Sciences Center in New Orleans, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Duke University, Durham, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Hamid Shah, MD, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas, Houston, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- University of Toronto/Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bak AB, Moghaddamjou A, Harrop JS, Aarabi B, Fehlings MG. The Impact of Interhospital Transfer on the Extent of Neurological Recovery in Acute Traumatic Spinal Cord Injury: Analysis of a Prospective Multicenter Data Set in 970 Cases. Neurosurgery. 2024 Jan 1;94(1):90-98. doi: 10.1227/neu.0000000000002642. Epub 2023 Aug 21. PMID 37607093
- See also: NACTN's Background, Mission, Sites and Resources — https://www.christopherreeve.org/research/nactn/about-nactn